CLINICAL TRIAL: NCT06782698
Title: Home-Based Physical Exercise During Neoadjuvant Treatment for Improving Fatigue and Quality of Life in Early Breast Cancer Patients (HoPEx-Breast): a Pragmatic Randomised Controlled Trial in a Portuguese Public Hospital
Brief Title: Home-Based Exercise Program During Neoadjuvant Treatment to Improve Fatigue and Quality of Life in Early HER2-Positive and Triple-Negative Breast Cancer Patients
Acronym: HoPEx-Breast
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário de Santo António (Other)
Collaborators: Oncology Research, Unit for Multidisciplinary Research in Biomedicine (UMIB), ICBAS-School of Medicine and Biomedical Sciences, University of Porto, Portugal (Unknown); Centro Hospitalar Universitário de Santo António, Unidade Local de Saúde de Santo António, Porto, Portugal (Unknown)
Responsible Party: Principal Investigator, Rita Carrilho Pichel, MD / PI, Centro Hospitalar Universitário de Santo António
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 002-24 DEFI 02 CE 02
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Triple Negative Breast Cancer (TNBC); HER2-Positive Breast Cancer; Early Breast Cancer; Cancer-related Fatigue; Quality of Life (QOL)
Keywords: Exercise; Home-based; Breast cancer; Fatigue; Quality of Life; Patient-reported outcomes; Physical activity; Neoadjuvant
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Masking Description: Pathologists who evaluate the pathological response are masked from the study-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based exercise program (Experimental): Participants allocated to the intervention arm will follow a home-based program, consisting of two initially supervised explanatory sessions, followed by home sessions of muscular training (twice per week), complemented with additional periods of aerobic exercise (20-30min trice per week). They will also receive routine short counseling for promotion of physical activity.
  Interventions: Behavioral: Home-based exercise program; Behavioral: Promotion of Healthy Physical Activity
- Short counselling for promotion of physical activity (Active Comparator): Participants allocated to the control arm will receive routine short counseling for promotion of physical activity, as recommended by the Portuguese Directorate-General of Health (Mendes R, et al. 2020)
  Interventions: Behavioral: Promotion of Healthy Physical Activity

INTERVENTIONS:
Behavioral: Home-based exercise program — The home-based program follows the National recommendations on Physical Exercise for Cancer Patients [Bruno RC, 2023]. It is logbook-guided and technology-enabled.
  It consists of:
  * Two initial supervised explanatory sessions, in the Physic and Rehabilitation Medicine Gym of our institution.
  * Followed by 2 muscular training sessions + 3 additional periods of aerobic exercise per week in their home environment until the end of neoadjuvant treatment. Patients are given a logbook with instructions and a sports bracelet for heart rate monitoring.
  The training sessions will be monitored by smartwatch heart rate measurements and self-notion of effort according to Borg Categorization [Borg GA, 1982] and recorded by the participants in the Mi Fitness application or an Exercise Diary.[Nilsen TS, 2018]
  Other Names: HoPEx-Breast intervention; Exercise
  Arms: Home-based exercise program
Behavioral: Promotion of Healthy Physical Activity — The short counseling consists of at least one opportunistic talk for promotion of physical activity, taking up to 5 minutes, during the Medical Oncology appointment or during Physical Assessments at T0. It should follow the instructions of the Portuguese Directorate-General of Health, "Short Counselling for the Promotion of Physical Activity", including the delivery of a Physical Activity Guide plus a Auxiliar of Decision or a Plan of Action or Maintenance.[Mendes R, 2020] All patients will receive a Guide about Nutrition for Cancer Patients [Capela AM, 2023] and may be offered Nutritional, Psychological or other additional consultations according to clinical judgement of the Medical Oncologist.
  Other Names: Short counseling; Control

SUMMARY:
The goal of this trial is to learn if a home-based exercise program (intervention) reduces fatigue and improves quality of life in adult patients with early breast cancer who are proposed for preoperative chemotherapy.

Conducted at Centro Hospitalar Universitário de Santo António, Porto, Portugal. It compares a structured exercise program prescribed by the physical and rehabilitation medicine team to routine counseling for physical activity by the medical oncologist.

All participants will:

1. Visit the hospital 3 times for physical assessments, at beginning of chemotherapy (T0), at 3-months (T1) and 1 month after surgery (T2)
2. Reply to questionnaires of fatigue and quality of life, at T0, T1 and T2
3. Adhere to routine medical oncology visits, treatments and exams

Participants of the intervention-arm will additionally:

1. Receive a exercise book, with exercise instructions and calendar
2. Have two in-person lessons about the exercise program
3. Visit the hospital 1 additional time, to have the second lesson
4. Wear a sport bracelet while exercising, to monitor heart rate Recruitment began in April 2024, with results to be shared in medical publications and conferences.

ELIGIBILITY:
Inclusion Criteria (must meet all):

* Adult patients,
* Any gender,
* Diagnosed with breast cancer, of HER2-positive or triple-negative subtypes,
* Proposed to neoadjuvant systemic cancer therapy. May be included: Patients non-eligible for anthracyclines or anti-HER2 therapies; patients with oligometastatic disease proposed for primary/neoadjuvant systemic cancer therapy with intent of radical treatment.

Exclusion Criteria:

* Patients that do not perform any neoadjuvant antineoplastic therapy, for example because of refusal, impeditive comorbidities, re-staging or other reasons.
* Contraindications for exercise or impediments to perform the intervention program, because of previous comorbidities or according to medical assessment (e.g. blindness).
* Patients who are unable to take questionnaires because of language or cognitive barriers (even with small help from a relative or investigator, still cannot answer properly).
* Luminal-like subtype, with hormonal receptor expression and HER2-negative.

Individual participants will be discontinued from the trial, in agreement with their physician where appropriate, if any health problem arises that will significantly affect their safety to participate in exercise for more than one month or if the participant decides to withdraw their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Changes in health-related quality of life, measured by EORTC QLQ-30, from baseline (T0) to 12 weeks of systemic therapy (T1) and to 1 month after surgery (T2)
Fatigue | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Changes in patient-reported fatigue, measured by FACIT-Fatigue, from baseline (T0) to 12 weeks of systemic therapy (T1) and to 1 month after surgery (T2)

SECONDARY OUTCOMES:
Exercise capacity | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Change on exercise capacity, measured as 6MWT distance, from T0 to T1 and from T0 to T2.
Physical activity levels | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Change on physical activity levels, measured by IPAQ-SF questionnaire (or by accelerometer), from T0 to T1 and from T0 to T2.
Hand grip strength | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Change on hand grip strength, from T0 to T1 and from T0 to T2.
Timed Up and Go | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Change on "Timed Up and Go", from T0 to T1 and from T0 to T2.
Complete pathologic response rate | From 1 month up to 2 months after breast surgery. Data can be restropectively collected from the pathologic report after this period.
  Percentage of participants of each arm that achieved complete pathological response, as assessed by a dedicated pathologist from our institution, blinded for the intervention.
Compliance to intervention | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Rate of participants that accepted to participate, that completed intervention, and the percentage of programed exercise sessions that were completed ", at T0, T1 and T2.
Safety | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Reported adverse events potentially related to exercise.
Compliance to questionnaires | From enrolement to up to 2 months after the end of intervention period, i.e. after breast surgery
  Rate of participants who replied to the quality of life and fatigue questionnaires, at T0, T1 and T2.

OTHER OUTCOMES:
Lymphedema | From enrolement to up to 12 months after the end of intervention period.
  Changes in arms circumferences from T0 to T2, and from T0 to 6-12m after the surgery.
Disease free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Time from the beginning of neoadjuvant treatment until death or recurrence of breast cancer disease.
Overall survival | From date of randomization until the date of death from any cause, assessed up to 120 months
  Time from the beginning of neoadjuvant treatment until death.
Health costs | From enrolement up to 6 months after surgery.
  Health costs estimation based on number of emergency episodes, in-hospital days, delayed day hospital sessions, off-labor days.

CONTACTS AND LOCATIONS:
Overall Officials: António Araújo, MD PhD, Study Director — Centro Hospitalar Universitário de Santo António, Unidade Local de Saúde de Santo António, Serviço de Oncologia Médica, Porto, Portugal. Oncology Research, UMIB, ICBAS-School of Medicine and Biomedical Sciences, University of Porto, Porto, Portugal.
Locations (1):
- Centro Hospitalar Universitário de Santo António, Unidade Local de Saúde de Santo António, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The anonymized individual participant data that will support the findings of this study will be available upon justified request to the corresponding author. The request will be analyzed by the research team and by the ethical and data protection committees of the institution.
Supporting Information: Study Protocol
Time Frame: From the registration of study and for five years after the closure of the study.